CLINICAL TRIAL: NCT06995001
Title: Phase I Study on the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of a Single Subcutaneous Injection of SHR-2173 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-2173-101
Record Dates: First submitted 2025-05-15; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treatment group A (Experimental)
  Interventions: Drug: SHR-2173
- Treatment group B (Experimental)
  Interventions: Drug: SHR-2173 ；Placebo
- Treatment group C (Experimental)
  Interventions: Drug: SHR-2173 ；Placebo
- Treatment group D (Experimental)
  Interventions: Drug: SHR-2173 ；Placebo
- Treatment group E (Experimental)
  Interventions: Drug: SHR-2173 ；Placebo

INTERVENTIONS:
Drug: SHR-2173 — SHR-2173 injection dose 1；
  Arms: Treatment group A
Drug: SHR-2173 ；Placebo — SHR-2173 injection dose 2 ；Pacebo dose 2
  Arms: Treatment group B
Drug: SHR-2173 ；Placebo — SHR-2173 injection dose 3 ；Pacebo dose 3
  Arms: Treatment group C
Drug: SHR-2173 ；Placebo — SHR-2173 injection dose 4 ；Pacebo dose 4
  Arms: Treatment group D
Drug: SHR-2173 ；Placebo — SHR-2173 injection dose 5 ；Pacebo dose 5
  Arms: Treatment group E

SUMMARY:
The study is being conducted to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics and immunogenicity of a single dose of SHR-2173 by subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female between the ages of 18 and 45 years, inclusive;
2. At least 50.0 kg for male subjects, 45.0 kg for female subjects, with a Body Mass Index (BMI) between 19.0-28.0 kg/m2 , inclusive (BMI = weight/height2 );
3. Female subjects of childbearing potential or male subjects whose partners are women of childbearing must avoid sperm/ovum donation and adopt highly effective contraceptive measurements (non-pharmacological contraception is required during the trial period) from the time of signing the informed consent form until the final visit;
4. Subjects who could understand the details, procedures, and possible adverse reactions of the trial before it begins and voluntarily sign a written informed consent form。

Exclusion Criteria:

1. Subjects with a history of drug allergies, or those with an allergic constitution (e.g., allergic to two or more drugs, foods, or pollens), or those known to be allergic to the investigational drug (including excipients) or similar drugs;
2. History or presence of any condition that may affect the safety or the pharmacokinetics of the investigational drug, including: immune system, respiratory system, hematological system (e.g., hemolytic reactions), circulatory system, digestive system, urinary system, nervous system, endocrine system, psychiatric disorders, metabolic disorders, or other conditions deemed unsuitable for participation in clinical trials;
3. Presence of active infection;
4. History of severe herpes virus infection, or history or presence of malignant tumors;
5. History of risk factors for torsades de pointes ventricular tachycardia, such as unexplained syncope, confirmed long QT syndrome (including family history), heart failure, myocardial infarction, or angina pectoris;
6. Subjects who have undergone major surgery within 3 months prior to screening, or surgery that may significantly affect the pharmacokinetics or safety evaluation of the investigational drug, or those planning to undergo surgery during the trial period.
7. Subjects who have used or are currently using any prescription drugs, over-the-counter medications, functional vitamins, health supplements, or herbal products within 2 weeks prior to dosing; or those planning to use other drugs during the trial period;
8. Subjects who have been vaccinated within 30 days prior to dosing or plan to be vaccinated within 3 months after dosing.
9. Subjects with a 12-lead ECG showing first-degree or higher atrioventricular block, atrial fibrillation or flutter, QTcF ≥450 ms, or other clinically significant abnormalities as judged by the investigator during the screening period;
10. Subjects with clinically significant abnormalities in blood routine, urinalysis, blood biochemistry, coagulation function, physical examination, vital signs, chest X-ray, or abdominal ultrasound as judged by the investigator during the screening period;
11. Subjects with positive results for hepatitis B surface antigen, hepatitis C virus antibody, Treponema pallidum antibody, or human immunodeficiency virus (HIV) during the screening period;
12. Pregnant or lactating females, or subjects with a positive serum pregnancy test;
13. Subjects with a positive tuberculosis infection screening test (interferon-gamma release assay, IGRA); IGRA includes but is not limited to QuantiFERON-TB Gold In-Tube (QFT-GIT) and T-SPOT.TB. If the IGRA result is indeterminate, retesting is allowed. Subjects with two indeterminate results will be considered positive.
14. Subjects who participated in other clinical trials and used investigational drugs within 3 months prior to dosing, or whose last study ended less than 5 half-lives or the duration of biological effects (whichever is longer);
15. Subjects who donated blood or lost ≥200 mL of blood (excluding menstrual blood loss in females) within 3 months prior to dosing, or received blood transfusions or blood products, or donated platelets within 2 weeks prior to dosing, or plan to donate blood during or within 3 months after the trial;
16. Subjects who frequently consumed alcohol (i.e., more than 14 standard units per week [1 standard unit = 14 g of alcohol, e.g., 360 mL beer, 45 mL of 40% spirits, or 150 mL wine]) within 3 months prior to dosing, or cannot abstain from alcohol during the trial period; or subjects with a positive breath alcohol test at baseline;
17. Subjects with a history of drug abuse or illicit drug use, or a positive drug abuse screening test at baseline;
18. Subjects who smoked more than 5 cigarettes or equivalent tobacco products daily within 3 months prior to dosing;
19. Subjects with abnormalities at the injection site, as judged by the investigator to be unsuitable for subcutaneous administration;
20. Any other reasons deemed unsuitable for participation by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2024-04-28 (Actual); Primary Completion 2024-11-28 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent Adverse Events (TEAE) | Day1~Day71

SECONDARY OUTCOMES:
Cmax | Day1~Day71
AUC0-t | Day1~Day71
AUC0-∞ | Day1~Day71
Tmax, | Day1~Day71
t1/2, | Day1~Day71
CLz/F, | Day1~Day71
Vz/F, | Day1~Day71
Immunogenicity ：Anti- SHR -2173 antibody (ADA) | Day1~Day71

CONTACTS AND LOCATIONS:
Locations (1):
- Haikou People's Hospital, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: Undecided